CLINICAL TRIAL: NCT04183647
Title: Investigation of Acute Effects of Local Vibration and Whole-Body Vibration Applications on Postural Control in Adult Patients With Ataxia
Brief Title: Investigation of Acute Effects of Local Vibration and Whole-Body Vibration Applications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, physical therapist, Hacettepe University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Vibration Applications
Record Dates: First submitted 2019-11-24; First posted 2019-12-03 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Ataxia
Keywords: local vibration, whole body vibration, postural control
MeSH Terms: conditions — Ataxia

STUDY DESIGN:
Intervention Model Description: Between the applications, a washout period of one week will be given to each patient to apply both local and whole body vibrations.
Who Masked: Outcomes Assessor
Masking Description: The study was planned as a single blind. Evaluations will be made by the blind evaluator.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local Vibration / Whole body vibration (Active Comparator): Local vibration will be sequentially applied to the bilateral gastrosoleus complex with the Vibrasens © device. Application, the largest part of the muscle, each limb 5'er for a total of 10 minutes, static semi-squat position will be done.
  The vibration frequency is 80 Hz and the amplitude is 1 mm.
  Interventions: Device: whole body vibration / local vibration
- Whole body vibration/local vibration (Active Comparator): Whole body vibration application will be done with Compex® Winplate device. During this application, patients will be asked to continue static semi-squat position with 5 minutes of vibration and then 5 minutes of vibration.Vibration frequency, 30 Hz amplitude will be selected 2 mm.
  Interventions: Device: whole body vibration / local vibration

INTERVENTIONS:
Device: whole body vibration / local vibration — Both the whole-body vibration application and the local vibration application will be applied to the patients in our cross-over study. Between the two applications will be given a washout period of one week. Patients will be evaluated both local and whole body vibration applications, 1 minute and 60 minutes after the end of the applications. After the evaluation, the patient will be rested in the sitting position until the evaluation at the 60th minute.

SUMMARY:
This study was designed as a single-blind, randomized and cross-over study to investigate and compare the acute effects of local vibration (LV) and whole-body vibration (WBV) applications on postural control in adult patients with ataxia.

The study will be included in patients aged 18-50 years, including ataxia diagnosed by the neurologist and able to walk independently. Patients with pregnancy status, epilepsy, spasticity, implant / endoprosthesis / pacemaker, benign paroxysmal positional vertigo, history of fracture in the last 6 months and other neurological diseases other than ataxia will not be included in the study. Between the applications, a washout period of one week will be given to each patient to apply both local and whole body vibrations. The order of application will be decided by the coin toss randomization method. Descriptive evaluations of the patients will be done with Mini-BESTest and Trunk Impairment Scale. Stability limits and postural sways (Bertec Balance Check ScreenerTM), gait time - distance characteristics (GAITRite), functional mobility skills (Timed Up and Go Test), and static balances (One Leg Stance Test) before, 1 minute after the application and 60 minutes after the application.

ELIGIBILITY:
Inclusion Criteria:

* Located in the 18-50 age range, diagnosed with ataxia by the neurologist, patients who can walk independently

Exclusion Criteria:

* Patients with pregnancy status, epilepsy, spasticity, implant / endoprosthesis / pacemaker, benign paroxysmal positional vertigo, history of fracture in the last 6 months, and other neurological disorders other than ataxia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Mini-BESTest | The application will be made immediately after the evaluations are completed within the same day (on average 45 min before application).
  It will be used for performance-oriented balance assessment. The test consists of 14 items and is evaluated on a score of 0-2. In the test, "0" indicates the lowest function level and "2 en indicates the highest function level.
Trunk Impairment Scale | The application will be made immediately after the evaluations are completed within the same day (on average 30 min before application).
  It will be used to evaluate trunk control. The scale has 17 items, 3 of which are static balance 10 are dynamic balance, 4 are stabilizer muscles. The total score that can be obtained is minimum "0 minimum and maximum" 23..
Limits of Stability and Postural Sways | change from baseline at 1 min and 60 min after applications.
  Bertec Balance Check Screener (Model BP5050) force platform system will be used. This force platform will measure stability limits in 4 directions (anterior, posterior, right, left) and postural sways in 4 different conditions (firm surface -eyes open, firm surface-eyes closed, foam surface-eyes open, foam surface-eyes closed).
Time-Distance Characteristics of the Gait | change from baseline at 1 min and 60 min after applications.
  GAITRite (CIR System INC. Clifton, NJ 07012) walkway system will be used. GAITRite; It is an electronic walkway which consists of portable carpet and sensors embedded on the carpet and transfers every foot contact to the computer when individuals walk on the carpet. With GAITRite, base of support (cm), velocity (cm / s) and cadence (steps / min) parameters will be evaluated.
Timed Up and Go Test | change from baseline at 1 min and 60 min after applications.
  It will be used to evaluate functional mobility.
One Leg Stance Test | change from baseline at 1 min and 60 min after applications.
  It will be used to evaluate static balance. For the right and left lower extremities, eyes will be opened and closed in two ways.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed KILINÇ, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozvar GB, Ayvat E, Kilinc M. Immediate Effects of Local Vibration and Whole-body Vibration on Postural Control in Patients with Ataxia: an Assessor-Blind, Cross-over randomized trial. Cerebellum. 2021 Feb;20(1):83-91. doi: 10.1007/s12311-020-01187-7. Epub 2020 Sep 3. PMID 32880847